CLINICAL TRIAL: NCT05727020
Title: Volatile Organic Compound Assessment in Pancreatic Ductal Adenocarcinoma (VAPOR 1 / BIORESOURCE)
Brief Title: Volatile Organic Compound Assessment in Pancreatic Ductal Adenocarcinoma
Acronym: VAPOR
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Pancreatic Cancer UK (Other); Imperial College Healthcare NHS Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); The Leeds Teaching Hospitals NHS Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Royal Surrey County Hospital NHS Foundation Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Swansea Bay University Health Board (Other); Dorset County Hospital NHS Foundation Trust (Other Government); North Tees and Hartlepool NHS Foundation Trust (Other); University Hospital Plymouth NHS Trust (Other); Barts & The London NHS Trust (Other); Milton Keynes University Hospital NHS Foundation Trust (Other Government); Buckinghamshire Healthcare NHS Trust (Other); Southern Health (Other)
Responsible Party: Sponsor
Other Study IDs: 22HH7787
Record Dates: First submitted 2023-01-23; First posted 2023-02-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer
Keywords: Volatile organic compounds (VOCs); Breath analysis; Volatolomics; Metabonomics / Lipidomics; Transcriptomics; Microbiome Analysis; Organoids; Immune profiling
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Breath, Saliva, Blood, Urine, Pancreatic tissue, Duodenal aspirate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- VAPOR 1 - PDAC (pancreatic ductal adenocarcinoma): 304 treatment-naive patients with histologically-confirmed* PDAC will be recruited to provide breath samples.
  *Patients that are due to undergo surgery for suspected PDAC (without pre-operative histological confirmation) may still be recruited despite the lack of pre-operative histological confirmation, assuming PDAC is subsequently confirmed within the resected specimen.
  Interventions: Diagnostic Test: Breath test
- VAPOR 1 - Control patients with benign pancreatic disorders: 257 patients with new-onset diabetes mellitus or chronic pancreatitis will be recruited to provide breath samples.
  New-onset diabetes is defined as: HbA1c≥48mmol/mol (6.5%), diagnosed within the preceding 6 months.
  Interventions: Diagnostic Test: Breath test
- VAPOR 1 - Control patients with non-specific GI symptoms and a normal pancreas: 257 patients with non-specific gastrointestinal symptoms but a radiologically-normal pancreas will be recruited to provide breath samples.
  Imaging to confirm a normal pancreas (CT / MRI / ultrasound) must have occurred within the preceding 12 months.
  Interventions: Diagnostic Test: Breath test
- VAPOR Bioresource - PDAC (pancreatic ductal adenocarcinoma): 96 treatment-naive patients with histologically-confirmed* PDAC will be recruited to provide samples of breath, saliva, blood, urine, pancreatic tissue and duodenal aspirate.
  *Patients that are due to undergo surgery for suspected PDAC (without pre-operative histological confirmation) may still be recruited despite the lack of pre-operative histological confirmation, assuming PDAC is subsequently confirmed within the resected specimen.
  Interventions: Diagnostic Test: Collection of matched samples of breath, biofluids and pancreatic tissue
- VAPOR Bioresource - Control patients with benign pancreatic disorders: 96 patients with benign pancreatic disorders (such as intraductal papillary mucinous neoplasms, pancreatic mucinous cystic neoplasms, chronic pancreatitis) will be recruited to provide samples of breath, saliva, blood, urine, pancreatic tissue and duodenal aspirate.
  Interventions: Diagnostic Test: Collection of matched samples of breath, biofluids and pancreatic tissue

INTERVENTIONS:
Diagnostic Test: Breath test — Patients must be fasted for a minimum of six hours prior to sample collection. For patients undergoing surgery or a procedure (e.g. endoscopy), breath samples must be obtained pre-operatively / prior to the administration of sedation, anaesthetic or other pharmacological agents.
  Groups: VAPOR 1 - Control patients with benign pancreatic disorders; VAPOR 1 - Control patients with non-specific GI symptoms and a normal pancreas; VAPOR 1 - PDAC (pancreatic ductal adenocarcinoma)
Diagnostic Test: Collection of matched samples of breath, biofluids and pancreatic tissue — In accordance with routine clinical practices, patients will be fasted for a minimum of six hours prior to surgery. Exhaled breath, saliva, blood and urine will be collected immediately prior to surgery (before induction of general anaesthesia). Pancreatic tissue samples and duodenal aspirate which will be collected upon resection of the pancreatic specimen.
  Groups: VAPOR Bioresource - Control patients with benign pancreatic disorders; VAPOR Bioresource - PDAC (pancreatic ductal adenocarcinoma)

SUMMARY:
Patients with early pancreatic cancer often have symptoms that could also be caused by many common benign conditions, or no symptoms at all. Jaundice, weight loss and pain are 'red flag' symptoms of pancreatic cancer that are linked to incurable disease. At the moment only patients with 'red flag' symptoms are urgently referred for diagnostic testing to find out if they have the cancer. As a result, late diagnosis is a common feature of pancreatic cancer. This leads to limited treatment options being available to patients by the time they are diagnosed, and ultimately results in poor survival rates.

There is a clear need to improve earlier detection of pancreatic cancer so that patients with pancreatic cancer can be identified earlier and faster, enabling them to start treatment more quickly.

The study team is developing a non-invasive breath test that detects small molecules called volatile organic compounds (VOCs) that may be altered by pancreatic cancers. For patients with non-specific symptoms, this test would help general practitioners (GPs) to identify those patients that may indeed have an underlying pancreatic cancer, who would benefit from referral for specialised pancreatic cancer tests.

DETAILED DESCRIPTION:
Bioresource study to identify pathways responsible for VOC production: A total of 192 patients will be recruited to provide samples to create a pancreatic biobank. This will be comprised of two groups, each containing 96 patients: (i) patients undergoing resection for pancreatic ductal adenocarcinoma (PDAC); (ii) control patients undergoing pancreatic resection for benign pancreatic disorders (e.g. intraductal papillary mucinous neoplasms, pancreatic mucinous cystic neoplasms, chronic pancreatitis). The following biosamples will be collected from each patient: breath, saliva, blood, urine, pancreatic tissue, duodenal aspirate. Collected samples will be stored in a biobank and will be utilised in a wide range of studies to investigate the mechanisms of VOC production in PDAC. The following analyses will be undertaken: volatolomics, metabonomics / lipidomics, metagenomics / microbiome analysis, transcriptomics, and culture experiments (to establish bacterial, immune and organoid cultures).

VAPOR 1 clinical study: Up to 813 patients will be recruited for the development of this non-invasive PDAC detection model. This will be comprised of three groups: (i) patients with PDAC; (ii) control patients with specified benign pancreatic disorders (new-onset diabetes mellitus, or chronic pancreatitis); (iii) control patients with non-specific gastrointestinal symptoms but a radiologically-normal pancreas. Participants will be required to fast for 6 hours prior to breath sampling. After rinsing their mouth with water, patients will be asked to provide breath samples by exhaling into single-use breath collection bags. Breath will be transferred using a precision pump into thermal desorption (TD) storage tubes. Breath samples will be analysed in accordance with existing quality-controlled processes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Adult patients ≥ 18 years old
* VAPOR 1: patients with either a) Histologically confirmed PDAC*; b) New-onset diabetes mellitus or chronic pancreatitis; or c) Non-specific gastrointestinal symptoms, but a radiologically-normal pancreas
* VAPOR Bioresource: patients undergoing pancreatic resection for a) Histologically confirmed PDAC*; or b) Benign pancreatic disorders e.g. intraductal papillary mucinous neoplasms, pancreatic mucinous cystic neoplasms, chronic pancreatitis

Note: *Patients undergoing surgery for suspected PDAC (without pre-operative histological confirmation) may be recruited assuming PDAC is confirmed within the resected specimen.

Exclusion Criteria:

* Patients who have already received chemotherapy, radiotherapy or surgery for their PDAC
* History of another cancer within the previous five years
* Previous upper gastrointestinal surgery
* Patients who are unable to provide a breath sample
* Pregnant women
* Patients unable to provide informed written consent
* VAPOR 1: Patients with active infection, receiving immunosuppressive medications or antibiotics within the preceding eight weeks
* VAPOR Bioresource: Patients receiving immunosuppressive medications within the preceding eight weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen in a hospital (secondary or tertiary level care) setting or at an NHS diabetes centre.
Sampling Method: Non-Probability Sample
Enrollment: 1005 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Levels of VOCs present in breath of subjects with PDAC and controls | 24 months
  Gas Chromatography-Mass Spectrometry (GC-MS) will be used to identify the levels (measured in parts per billion, ppb) of certain cancer-associated VOCs in breath

SECONDARY OUTCOMES:
Levels of volatile metabolites present in headspace of the urine of subjects with PDAC and controls | 24 months
  Headspace sampling techniques will be used for headspace collection from urine samples. GC-MS will be used to determine the levels (measured in parts per billion, ppb) of certain cancer-associated VOCs within the headspace of urine.
Characterisation of bacterial species in saliva samples, pancreatic tissue samples and duodenal aspirate samples of subjects with PDAC compared to controls | 24 months
  Bacterial species present will be identified (measured) using sequencing techniques such as 16s or whole genome sequencing.
  * Bacteria within the saliva samples will be cultured and species isolated
  * Bacteria from pancreatic biopsies will be separated from the tissue, and will be cultured to isolate the bacterial species
  * Bacteria derived from duodenal aspirate will be cultured and species isolated
Levels of VOCs produced by the bacteria isolated from saliva samples, pancreatic tissue samples and duodenal aspirate samples of subjects with PDAC | 24 months
  The cancer-associated bacterial species isolated and identified as part of Outcome Measure 3 will then be re-cultured within a controlled environment. Headspace and media sampling will be performed to identify and measure the levels of volatile metabolites (measured in parts per billion, ppb) present using GC-MS and LC-MS (Liquid Chromatography-Mass Spectrometry) techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Professor George B Hanna, PhD, FRCS, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walsh CM, Murray J, Laponogov I, Parker A, Ellis JK, Converso V, Austin E, Boshier PR, Czajkowski C, Spalding D, Al-Mukhtar A, Frampton AE, Roberts KJ, Pandanaboyana S, Halloran C, Costello E, Kocher H, Mitra V, Hamady Z, Al-Sarireh B, Pathak S, Mitchell WK, Siriwardena AK, Westlake C, Pereira SP, Spiliotis I, Biswas S, Vapor Collaborators, Spanel P, Veselkov K, Sharples LD, Hanna GB; VAPOR Collaborators. Development and validation of a diagnostic prediction model for pancreatic ductal adenocarcinoma: VAPOR 1, protocol for a prospective multicentre case-control study. BMJ Open. 2025 Aug 27;15(8):e094505. doi: 10.1136/bmjopen-2024-094505. PMID 40866056